CLINICAL TRIAL: NCT03560986
Title: Placebo-controlled Efficacy and Safety Trial of Intravenous Neridronic Acid in Subjects With Complex Regional Pain Syndrome (CRPS)
Brief Title: Efficacy and Safety of Intravenous Neridronic Acid in Complex Regional Pain Syndrome (CRPS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KF7013-04; 2017-004244-37 (EudraCT Number); U1111-1203-5020 (Other: World Health Organization)
Record Dates: First submitted 2018-05-07; First posted 2018-06-19 (Actual); Results first posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Complex Regional Pain Syndrome (CRPS)
Keywords: Neridronic Acid; Neridronate; CRPS; Reflex sympathetic dystrophy (RSD)
MeSH Terms: conditions — Complex Regional Pain Syndromes; Reflex Sympathetic Dystrophy | interventions — 6-amino-1-hydroxyhexane-1,1-diphosphonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded treatment in Treatment Period A, open-label infusion in Treatment Period B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neridronic acid (Experimental): Neridronic acid 100 mg - 4 intravenous (i.v.) infusions within 10 days (i.e., on Days 1, 4, 7, and 10). The investigational medicinal product (IMP) was diluted in sterile normal saline to a volume of approximately 500 mL before slow administration.
  The maximum neridronic acid dose was 800 mg: 400 mg in Treatment Period A and 400 mg in Treatment Period B.
  Interventions: Drug: Neridronic acid 100 mg
- Placebo (Placebo Comparator): Matching placebo - 4 intravenous infusions within 10 days (i.e., on Days 1, 4, 7, and 10). The IMP was diluted in sterile normal saline to a volume of approximately 500 mL before slow administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neridronic acid 100 mg — 100 mg neridronic acid supplied in glass vials in 8 mL of excipients.
  Arms: Neridronic acid
Drug: Placebo — Glass vials with matching placebo.
  Arms: Placebo

SUMMARY:
The aim of this trial was to investigate the efficacy and safety of intravenous neridronic acid in subjects with Complex Regional Pain Syndrome (CRPS).

The trial consisted of an Enrollment Period lasting up to 60 days, Treatment Period A consisting of 4 infusions (neridronic acid 100 mg or placebo) over 10 days, and a Follow-up Period 1 until Week 26. At Week 26, participants meeting the pre-specified criteria entered the open-label Treatment Period B with 4 additional infusions (neridronic acid) over 10 days and follow-up visits until Week 52. Participants not meeting the pre-specified criteria to continue into Treatment Period B continued in Follow-up Period 2 until Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed.
* Male or female participant at least 18 years of age at Visit 1.
* A diagnosis of CRPS according to the clinical diagnostic criteria recommended by the International Association for the Study of Pain (IASP; "Budapest clinical criteria"), assessed at Visit 1. Signs and symptoms of CRPS must apply to an affected limb (arm or leg) and must demonstrate asymmetry with respect to the contralateral limb. The CRPS duration must be 2 years or less since onset of symptoms.
* A baseline average pain intensity score of greater than or equal to 4 using an 11-point numerical rating scale (NRS), referring to the CRPS-affected limb (average of pain recorded over 7 days). The baseline average pain intensity score will be calculated automatically by the electronic diary, which must be checked prior to allocation at Visit 2. A participant who has not met average baseline pain intensity requirements (at least 4 average pain intensity ratings) due to lack of compliance with the electronic diary may be rescheduled for Visit 2 (1 time only), with appropriate re-training to ensure compliance with use of the electronic diary.
* In stable treatment and follow-up therapy for CRPS for at least 1 month prior to allocation to treatment (Visit 2). Participants must have failed attempts with at least 2 available treatments for CRPS, 1 of which must have been a pharmacologic treatment.
* Women of child-bearing potential must have a negative urine Beta-human chorionic gonadotropin (ß-HCG) pregnancy test at Visit 1 and must be using 2 forms of medically acceptable contraception, including at least 1 highly effective method of contraception with a low failure rate, defined as less than 1% per year, and a second medically acceptable method such as use of condoms with spermicide by their male partner. A barrier method alone is not acceptable. Highly effective methods of contraception must be used for at least 1 month prior to Visit 2 and for the duration of the trial. Male participants must use condom and spermicide during intercourse and must take care that the female sexual partner uses at least 1 additional method of contraception with a low failure rate defined as above, starting with Visit 2 until at least 4 weeks after the last Investigational medicinal product (IMP) infusion.
* Participants must be able to communicate meaningfully, be able to differentiate with regard to location and intensity of the pain, and be able to answer the questions in the questionnaires used in this trial (assistance in filling out the questionnaires may be provided, if required due to motor or other physical impairment).

Exclusion Criteria:

* Evidence of renal impairment (estimated Glomerular Filtration Rate [eGFR] less than 30 mL/min/1.73 m2 using the 2009 Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] creatinine equation [Levey et al. 2009] or a urinary albumin to creatinine ratio [ACR] greater than 150 mg/g), based on central safety laboratory data obtained prior to Visit 2. Note: a single repeat laboratory test is allowed.
* Serum calcium or magnesium outside of the central laboratory's reference range, based on central safety laboratory data obtained prior to Visit 2 (a single repeat laboratory test is allowed); a history of hypocalcemia or a metabolic disorder anticipated to increase risk for hypocalcemia (e.g., hypoparathyroidism); anticipated need for any new drug with known potential to cause hypocalcemia (e.g., aminoglycosides, new treatment with or dose adjustment of loop diuretics) during the trial. Participants on a stable dose of loop diuretics may receive treatment with IMP as long as no dosage increases in the diuretic medication are anticipated and calcium levels are in the reference range.
* Vitamin D deficiency, defined as a 25(OH)D level less than 30 ng/mL (75 nmol/L), based on central safety laboratory data obtained prior to Visit 2 (up to 4 repeat laboratory tests are allowed). Participants with vitamin D deficiency should receive appropriate supplementation during the Enrollment Period. A vitamin D level of at least 30 ng/mL (75 nmol/L) must be documented prior to allocation to IMP.
* Corrected QT interval (according to Fridericia's formula; QTcF) greater than 470 ms (average of 3 Electrocardiogram (ECGs) obtained at Visit 1) according to central ECG reading facility evaluation or QTcF greater than 470 ms at pre-dose ECG at Visit 2 according to the investigator's judgment; serum potassium outside the central laboratory's reference range at Visit 1(a single repeat laboratory test is allowed); clinically unstable cardiac disease, including: unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia, or an indwelling pacemaker; evidence of complete left bundle branch block; complete atrioventricular block; history of Long QT Syndrome or a relative with this condition; or any history of or other known risk factor for torsade de pointes.
* Participants receiving medications with a known risk of torsades de pointes within 7 days prior to allocation. Participants receiving selective serotonin re-uptake inhibitor antidepressants are eligible if the QT interval values do not meet the exclusion criteria, the medication was started at least 1 month prior to allocation, the dose is stable, and the dose is anticipated to remain stable throughout the trial.
* Any prior use of a bisphosphonate for treatment of CRPS, any prior administration of a bisphosphonate within the previous year, anticipated requirement for treatment with a bisphosphonate for another condition such as osteoporosis during the trial, or administration of denosumab (Prolia®) or other bone turnover suppressing drugs within 6 months prior to Visit 1.
* History of any allergic or hypersensitivity reaction to neridronic acid or other bisphosphonate, acetaminophen, or to vitamin D or calcium supplements.
* Recent tooth extraction or other invasive dental procedure (within 3 months prior to Visit 1), unhealed or infected extraction site, or significant dental/periodontal disease that may pre-dispose to need for tooth extraction or other invasive dental procedures during the trial. Participants with indeterminate, suspicious or unreliable dental history, in the opinion of the investigator, must undergo a dental examination prior to receiving treatment.
* Evidence of denture-related gum trauma or improperly fitting dentures causing injury.
* Prior radiation therapy of the head or neck (within 1 year of Visit 1).
* History of malignancy within 2 years prior to Visit 1, with the exception of basal cell carcinoma.
* Use of nerve blocks, ketamine infusions, intravenous immunoglobulin, acupuncture, electromagnetic field treatment, or initiation/implementation of radiofrequency ablation or other sympathectomy procedures, or peripheral nerve stimulation within 6 weeks prior to Visit 1.
* Evidence of current alcohol or drug abuse, or history of alcohol or drug abuse within 2 years of Visit 1, based on participant history and physical examination and according to the investigator's judgment.
* Any other severe medical condition, including severe depression, or any other severe mood disorder, that in the opinion of the investigator may affect efficacy or safety assessments or may compromise the participants safety during trial participation.
* Women who are pregnant or breastfeeding.
* Elevated aspartate aminotransferase or alanine aminotransferase greater than 2-fold upper limit of normal, based on central safety laboratory data obtained at Visit 1, or current evidence of chronic liver disease. Safety laboratory testing may be repeated prior to Visit 2, and participants will be allowed in the trial if results of 2 consecutive tests, at least 3 days apart, are less than or equal to 2-fold upper limit of normal.
* Participation in another investigational drug trial within 3 months prior to Visit 1, or any previous trial involving neridronic acid, with the exception of participants participating in study KF7013-01 who were assigned to placebo and did not receive neridronic acid.
* Participant is engaged in litigation related to their disability from CRPS in which monetary gain or loss (or other compensation) may affect their objective participation in the trial.
* Participants taking forbidden concomitant medications/therapies or not being able to follow the rules of use of concomitant treatment.
* Participants incapable of giving informed consent.

Criteria to continue into Treatment Period B

* A value of at least 4 on the pain intensity question (question number 29, GLOBAL07) of the Patient-Reported Outcomes Measurement Information System (PROMIS®) (PROMIS-29 profile) at Visit 11.
* The following exclusion criteria are not met:

  * Evidence of renal impairment (eGFR less than 30 mL/min/1.73 m2 using the 2009 CKD-EPI creatinine equation [Levey et al. 2009] or a urinary ACR greater than 150 mg/g), based on central safety laboratory data obtained prior to Visit 11. A single repeat laboratory test is allowed.
  * Corrected QT interval (QTcF) greater than 470 ms (average of 3 ECGs obtained at Visit 10) according to the central ECG reading facility evaluation or QTcF greater than 470 ms at pre-dose ECG at Visit 11 according to the investigator's judgment; serum potassium outside the central laboratory's reference range at Visit 10 (a single repeat laboratory test is allowed); clinically unstable cardiac disease, including: unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia, or an indwelling pacemaker; evidence of complete left bundle branch block; complete atrioventricular block; any other known risk factor for torsade de pointes.
  * Participants receiving medications with a known risk of torsades de pointes within 7 days prior to re-allocation.
  * Participants taking forbidden concomitant medications/therapies or not being able to follow the rules of use of concomitant treatment.
  * Recent tooth extraction or other invasive dental procedure (within 3 months prior to Visit 11), unhealed or infected extraction site, or significant dental/periodontal disease that may pre-dispose to need for tooth extraction or other invasive dental procedures during the further course of the trial.
  * Serum calcium outside of the central laboratory's reference range, despite appropriate supplementation between Visit 10 and Visit 11, based on the last central safety laboratory data obtained prior to Visit 11. Two repeat laboratory tests are allowed.
  * Vitamin D deficiency prior to IMP re-allocation, defined as a 25(OH)D level less than 30 ng/mL (75 nmol/L), based on the last central safety laboratory data obtained prior to Visit 11, i.e., inability to normalize 25(OH)D levels to at least 30 ng/mL (75 nmol/L) despite appropriate supplementation between Visit 10 and Visit 11. Two repeat laboratory tests are allowed.
  * Elevated aspartate aminotransferase or alanine aminotransferase greater than 2-fold upper limit of normal, based on central safety laboratory data obtained at Visit 10, or current evidence of chronic liver disease. A single repeat laboratory test is allowed.
* No other criterion for trial and/or IMP discontinuation is met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (71):
- United States (41):
  - US446 - Clinical Trial Connection, Cottonwood, Arizona
  - US453 - Physicians Research Group II, LLC, Tempe, Arizona
  - US428 - Quality of Life Medical and Research Center LLC, Tucson, Arizona
  - US422 - Woodland International Research Group, Little Rock, Arkansas
  - US454 - Alliance Research Institute, Canoga Park, California
  - US415 - Clearview Medical Research LLC, Canyon Country, California
  - US410 - Alliance Research Centers, Laguna Hills, California
  - US432 - Torrance Clinical Research Institute Inc., Lomita, California
  - Us414 - Alexander Ford Md, Los Angeles, California
  - US441 - Samaritan Center for Medical Research, Los Gatos, California
  - US406 - CI Trials, Santa Ana, California
  - US411 - Syrentis Clinical Research, Santa Ana, California
  - US420 - Mountain View Clinical Research, INC, Denver, Colorado
  - US447 - ASCLEPES Research Centers, Brooksville, Florida
  - US457 - Florida Spine Institute, Clearwater, Florida
  - US430 - South Lake Pain Institute, Clermont, Florida
  - US434 - Finlay Medical Research, Miami, Florida
  - US407 - Oceane 7 Medical and Research Center, Inc., Miami, Florida
  - US436 - Cordova Research Institute, Miami, Florida
  - US417 - Tampa Pain Relief Center, Tampa, Florida
  - US403 - Palm Beach Research Center, West Palm Beach, Florida
  - US404 - Infinite Clinical Trials, Riverdale, Georgia
  - US424 - Georgia Neurology and Sleep Medicine Assoc., Suwanee, Georgia
  - US431 - Injury Care Research, LLC, Boise, Idaho
  - US437 - Great Lakes Clinical Trials LLC, Chicago, Illinois
  - US435 - Centex Studies Inc, Lake Charles, Louisiana
  - US448 - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - US450 - SRI International, Plymouth, Michigan
  - US449 - Michigan Pain Consultants, Wyoming, Michigan
  - US433 - Creighton University - Osteoporosis Research Center, Omaha, Nebraska
  - US419 - Manhattan Behavioral Medicine, New York, New York
  - US440 - OnSite Clinical Solutions LLC, Charlotte, North Carolina
  - US405 - OnSite Clinical Solutions LLC, Hickory, North Carolina
  - US416 - Medical Research International, Oklahoma City, Oklahoma
  - US429 - Lehigh Valley Health, Allentown, Pennsylvania
  - US438 - Abington Neurological Associates, LTD., Willow Grove, Pennsylvania
  - US425 - PCPMG Clinical Research Unit LLC, Greenville, South Carolina
  - US423 - Biopharma Informatic Inc. Research Center, Houston, Texas
  - US443 - Centex Studies Inc, Houston, Texas
  - US421 - Northwest Clinical Research Center, Bellevue, Washington
  - US445 - Exemplar Research Inc, Morgantown, West Virginia
- Canada (6):
  - CA404 - Jeffrey Weinberg Medicine Professional Corporation c/o Jacobs Pain Center, Markham, Ontario
  - CA406 - Malton Medical Centre (attn: Vrijender Singh), Mississauga, Ontario
  - CA402 - SKDS Research Inc, Newmarket, Ontario
  - CA407 - King Street Medical Clinic, Oshawa, Ontario
  - CA403 - Bluewater Clinical Research Group, Sarnia, Ontario
  - CA405 - Canadian Centre for Clinical TrialsCCCT, Thornhill, Ontario
- Czechia (3):
  - CZ403 - CCBR Ostrava, Ostrava
  - CZ402 - CCR Czech a,s., Pardubice
  - CZ401 - FORBELI s.r.o., Prague
- Poland (3):
  - PL405 - Medical Solutions, Elblag
  - PL404 - Zagiel Med Sp Zoo, Lublin
  - PL403 - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp.z o.o, Tarnów
- Serbia (4):
  - RS401 - Clinical Center of Serbia, Clinic for physical medicine and rehabilitation, Belgrade
  - RS403 - Clinical Center Kragujevac, Department of Physical Medicine and rehabilitation, Kragujevac
  - RS404 - Clinical Center Nis, Clinic for Physical Medicine and Rehabilitation, Niš
  - RS405 - Clinical Center of Vojvodina, Medical Rehabilitation Clinic, Novi Sad
- Slovakia (4):
  - SK402 - MUDr. Beata Dupejova, neurologicka ambulancia sro, Banská Bystrica
  - SK404 - Medical Center Konzilium, Dubnica nad Váhom
  - SK403 - NEURES, s.r.o., Krompachy
  - SK401 - MUDr. Viliam Cíbik, PhD, Algeziologická ambulancia, Pruské
- United Kingdom (10):
  - GB413 - MAC Clinical Research, Barnsley
  - GB412 - MAC Clinical Research, Blackpool
  - GB415 - MAC Clinical Research, Cannock
  - GB416 - Royal Devon and Exeter Hospital, Exeter
  - GB410 - MAC Clinical Research, Leeds
  - GB409 - MAC Clinical Research, Liverpool
  - GB407 - Pain and Neuromodulation Centre Ground Floor, Gassiot House, St Thomas Hospital, London
  - GB402 - St Pancras Clinical Research, London
  - GB408 - MAC Clinical Research, Manchester
  - GB414 - MAC Clinical Research, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Group Web Site (see URL below for details); according to the European Federation of Pharmaceutical Industries and Associations (EFPIA) Data Sharing Principles.
Supporting Information: Study Protocol, SAP
URL: http://www.grunenthal.com/r-d-vision-mission/clinical-trials/data-sharing-clinical-trials

REFERENCES:
- [Background] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrollment on 31 May 2018. After a pooled interim analysis of primary endpoint data of studies KF7013-04 and KF7013-02 (NCT03530345), recruitment was stopped as interim results indicated futility. Last participant's last assessment was on 01 Aug 2019.
Pre-assignment Details: 267 participants were enrolled (signed consent), 100 were allocated to treatment, and 99 received study medication. Of 167 participants not allocated, 99 did not meet inclusion/met exclusion criteria, 3 were lost to follow-up, 14 withdrew consent, 1 experienced adverse events, and 50 were not allocated for other reasons (study termination).
Groups:
- Neridronic Acid - Treatment Period A: * Treatment Period A: Neridronic acid 100 mg - 4 intravenous infusions within 10 days; Follow-up Period 1 until 26 weeks.
  * Treatment Period B: Neridronic acid 100 mg - 4 intravenous infusions within 10 days; Follow-up Period 2 until 52 weeks.
- Placebo - Treatment Period A: * Treatment Period A: Matching placebo - 4 intravenous infusions within 10 days; Follow-up Period 1 until 26 weeks.
  * Treatment Period B: Neridronic acid 100 mg - 4 intravenous infusions within 10 days; Follow-up Period 2 until 52 weeks.
Period: Treatment Period A/Follow-up Period 1
Arm/Group | Neridronic Acid - Treatment Period A | Placebo - Treatment Period A
Started | 48 | 51 (One additional participant was allocated to placebo but not treated.)
Treatment Period A Completers | 45 | 45
Completed (Participants completing Follow-up Period 1.) | 12 | 13
Not Completed | 36 | 38
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Disc. before end of Follow-up Period 1 | 32 | 35
Period: Treatment Period B/Follow-up Period 2
Arm/Group | Neridronic Acid - Treatment Period A | Placebo - Treatment Period A
Started | 9 (3 Participants completed Treatment Period A/Follow-up Period 1 but were not allocated in Period B.) | 8 (5 Part. completed Placebo Treatment Period A/Follow-up Period 1 but were not allocated in Period B.)
Treatment Period B Completers | 8 | 8
Completed (Participants completing Follow-up Period 2.) | 1 | 0
Not Completed | 8 | 8
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Disc. before end of Follow-up Period 2 | 7 | 7

BASELINE CHARACTERISTICS:
Population: Safety Set; all participants treated in Treatment Period A.
Groups:
- Neridronic Acid - Treatment Period A: Neridronic acid 400 mg administered by 4 intravenous infusions within 10 Days in Treatment Period A.
- Placebo - Treatment Period A: Matching placebo administered by 4 intravenous infusions within 10 Days in Treatment Period A.
- Total: Total of all reporting groups
Arm/Group | Neridronic Acid - Treatment Period A | Placebo - Treatment Period A | Total
Number analyzed (Participants) | 48 | 51 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (12.7) | 50.4 (12.6) | 50.0 (12.6)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0
  From 18 to <65 years | 42 | 46 | 88
  From 65 to <85 years | 6 | 5 | 11
  85 years and above | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 13 | 15 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 42 | 44 | 86
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1 | 4 | 5
  United States | 37 | 36 | 73
  Czechia | 5 | 4 | 9
  United Kingdom | 2 | 5 | 7
  Slovakia | 3 | 2 | 5
CRPS type [Count of Participants; unit: Participants] — CRPS Type I: Occurs after a minor or major tissue injury without clinical signs of major peripheral nerve injury.
  CRPS Type II: Occurs after an injury with clinical signs of major peripheral nerve injury.
  Participants
    CRPS Type I | 38 | 33 | 71
    CRPS Type II | 5 | 9 | 14
    Unknown CRPS Type | 5 | 9 | 14
Time since onset of CRPS symptoms [Median (Inter-Quartile Range); unit: months] | 12.88 [7.30 to 18.90] | 11.80 [6.00 to 18.57] | 12.33 [6.63 to 18.57]
Time since diagnosis of CRPS [Median (Inter-Quartile Range); unit: months] | 5.92 [0.87 to 11.03] | 5.83 [0.03 to 15.03] | 5.83 [0.47 to 12.63]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Average Pain Intensity Score (Weekly Average of Pain Values Recorded Daily in the Electronic Diary)
Description: In the Baseline Phase and in Treatment Period A/Follow-up Period 1, participants were asked to assessed their average CRPS-related pain on an 11-point numerical rating scale (NRS) - from 0 = "no pain" to 10 = "pain as bad as you can imagine" and report it once daily (in the evening, 24-hour recall) in an electronic diary.
  Changes from baseline (average for the Baseline Phase) to the weekly average for Week 12 were calculated.
Time Frame: From the Baseline Phase (Day -7 to Day -1) to Week 12
Population: Full Analysis Set; all participants treated in Treatment Period A with all data available at the time of last participant out following premature study termination.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Neridronic Acid - Treatment Period A: Neridronic acid 100 mg - 4 intravenous infusions within 10 Days
- Placebo - Treatment Period A: Matching placebo - 4 intravenous infusions within 10 Days
Arm/Group | Neridronic Acid - Treatment Period A | Placebo - Treatment Period A
Number analyzed (Participants) | 48 | 51
units on a scale | -1.28 (0.270) | -1.71 (0.268)
Statistical Analysis 1: Comparison: Neridronic Acid - Treatment Period A vs Placebo - Treatment Period A; Mixed-effects model for repeated measures (MMRM) defined with baseline pain intensity as covariate, the factors geographic region, week, treatment and treatment-by-week as fixed effects, and an unstructured covariance matrix to model the covariance structure of the repeated measurements; Test type: Superiority; p = 0.2522, Mixed Models Analysis — 2-sided p-value for testing superiority of neridronic acid 400 mg compared to placebo; The degrees of freedom of the denominator are estimated using the Kenward-Roger approximation; Mean Difference (Net) = 0.43, 95% CI 2-sided [-0.31 to 1.17], Standard Error of Mean 0.372 — The primary endpoint estimate was the least squares mean differences of change from baseline in pain NRS (electronic diary) at Week 12 between neridronate and Placebo

2. Secondary Outcome: Change From Baseline to Week 26 in the Average Pain Intensity Recorded on the Tablet Computer
Description: 11-point NRS - from 0 = "no pain" to 10 = "pain as bad as you can imagine" - reported at the visits on a tablet computer (24-hour recall). Changes from baseline to Week 26 were planned to be analyzed.
Time Frame: From baseline (Visit 2 [Day 1]) to Visit 11 (Week 26)
Population: Data were not collected or analyzed because a confirmatory testing strategy was not performed as pre-specified in the protocol that secondary endpoints would only be tested if neridronic acid was superior to placebo on the primary outcome measure. A confirmatory or descriptive analysis was not performed due to early study termination.
Arm/Group | Neridronic Acid - Treatment Period A | Placebo - Treatment Period A
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pain Response to Treatment, Defined as at Least 30% Decrease From Baseline in the Average Pain Intensity at Week 12, Recorded on the Tablet Computer
Description: 11-point NRS - from 0 = "no pain" to 10 = "pain as bad as you can imagine" - reported at the visits on a tablet computer (24-hour recall).
  The number of participants with response at Week 12 was planned to be determined.
Time Frame: From baseline (Visit 2 [Day 1]) to Visit 8 (Week 12)
Population: as for outcome 2
Arm/Group | Neridronic Acid - Treatment Period A | Placebo - Treatment Period A
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pain Response to Treatment, Defined as at Least 30% Decrease From Baseline in the Average Pain Intensity at Week 26, Recorded on the Tablet Computer
Description: 11-point NRS - from 0 = "no pain" to 10 = "pain as bad as you can imagine" - reported at the visits on a tablet computer (24-hour recall). The number of participants with response at Week 26 was planned to be determined.
Time Frame: From baseline (Visit 2 [Day 1]) to Visit 11 (Week 26)
Population: as for outcome 2
Arm/Group | Neridronic Acid - Treatment Period A | Placebo - Treatment Period A
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline to Week 12 in the Pain Intensity Level of Dynamic Mechanical Allodynia (DMA)
Description: Dynamic mechanical allodynia: a tactile stimulus is applied in a single sweeping motion (1 cm to 2 cm length) on the skin on the affected limb. The participants are asked to judge the stimulus intensity by means of an NRS (0 to 10). "0" in this case means "no pain". Each "pricking", "stinging" or "burning" sensation is defined as a painful sensation, which should always be evaluated by giving a value greater than "0". "10" corresponds to the individual maximum pain imaginable. Change from baseline was planned to analyzed.
Time Frame: From baseline (Visit 2 [Day 1]) to Visit 8 (Week 12)
Population: as for outcome 2
Arm/Group | Neridronic Acid - Treatment Period A | Placebo - Treatment Period A
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline to Week 12 in the Pressure Pain Threshold (PPT) Ratio for the Thenar Muscle/Abductor Hallucis Muscle
Description: Pressure pain threshold: using a pressure algometer (contact area 1 cm2), the threshold for pressure-induced pain is measured on the thenar muscle/abductor hallucis muscle in 3 series of slowly increasing stimulus intensities (at a rate of about 50 kPa/s). The threshold is then determined as the arithmetic mean of the 3 series (in kPa).
  The ratio of the thresholds of the affected limb versus the unaffected limb was planned to be calculated.
Time Frame: From baseline (Visit 2 [Day 1]) to Visit 8 (Week 12)
Population: as for outcome 2
Arm/Group | Neridronic Acid - Treatment Period A | Placebo - Treatment Period A
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline to Week 12 in the Ratio of the Figure of Eight Measurements of the Affected Limb Versus the Unaffected Limb
Description: In participants with the CRPS sign of edema on the CRPS severity score at baseline, circumference of the hand or foot will be measured by the investigator with measurement tape using the figure-of-eight method at both the affected limb and the contralateral unaffected limb. Each measurement will be performed 3 times. The average of the 3 measurements will be used for further analysis.
  The ratio of the averages of the affected limb versus the unaffected limb was planned to be calculated and used for the determination of the change from baseline.
Time Frame: From baseline (Visit 2 [Day 1]) to Visit 8 (Week 12)
Population: as for outcome 2
Arm/Group | Neridronic Acid - Treatment Period A | Placebo - Treatment Period A
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were documented from the time of enrollment (i.e., the time the informed consent form was signed) up to the time of the last protocol scheduled contact, i.e., date of last visit/contact (could be a phone call, e.g., in case of withdrawal). Only treatment emergent adverse events (TEAEs, i.e., those reported from baseline (after first administration of study medication) are reported in the tables below.
Description: Participants with TEAEs may be presented in 2 of 6 reporting groups depending on the time the TEAEs were reported.
  * Treatment Period A/Follow-up Period 1 (TPA): Baseline to Week 26 (Placebo or neridronic acid).
  * Treatment Period B/Follow-up Period 2 (TPB): Week 26 to Week 52 (follow-up without study medication administration) or Week 26 to Week 52 (participants with neridronic acid treatment after placebo and those receiving re-treatment with neridronic acid).
Groups:
- Baseline to Week 26: Placebo TPA: In Treatment Period A, participants received matching placebo - 4 intravenous infusions within 10 Days; Follow-up Period 1 until 26 weeks.
- Baseline to Week 26: Neridronic Acid TPA: In Treatment Period A, participants received neridronic acid 100 mg - 4 intravenous infusions within 10 days; Follow-up Period 1 until 26 weeks.
- Week 26 to Week 52: Placebo TPA: Participants with placebo treatment in Treatment Period A/Follow-up Period 1 were followed up without administration of study medication until 52 weeks in Follow-up Period 2.
- Week 26 to Week 52: Placebo TPA, Neridronic Acid TPB: Participants who had completed treatment with placebo in Treatment Period A/Follow-up Period 1 received neridronic acid treatment (100 mg - 4 intravenous infusions within 10 days) in Treatment Period B/Follow-up Period 2 until 52 weeks.
- Week 26 to Week 52: Neridronic Acid TPA: Participants who had completed treatment with neridronic acid treatment in Treatment Period A/Follow-up Period 1 were followed up without administration of study medication until 52 weeks in Follow-up Period 2.
- Week 26 to Week 52: Neridronic Acid TPA, Neridronic Acid TPB: Participants who had completed treatment with neridronic acid in Treatment Period A/Follow-up Period 1 received re-treatment with neridronic acid 100 mg - 4 intravenous infusions within 10 days; Follow-up Period 2 until 52 weeks.
Arm/Group | Baseline to Week 26: Placebo TPA | Baseline to Week 26: Neridronic Acid TPA | Week 26 to Week 52: Placebo TPA | Week 26 to Week 52: Placebo TPA, Neridronic Acid TPB | Week 26 to Week 52: Neridronic Acid TPA | Week 26 to Week 52: Neridronic Acid TPA, Neridronic Acid TPB
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/48 | 0/43 | 0/8 | 0/39 | 0/9
Serious Adverse Events (participants affected / at risk) | 3/51 | 2/48 | 0/43 | 1/8 | 0/39 | 1/9
Other Adverse Events (participants affected / at risk) | 40/51 | 40/48 | 1/43 | 6/8 | 0/39 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline to Week 26: Placebo TPA (N=51) | Baseline to Week 26: Neridronic Acid TPA (N=48) | Week 26 to Week 52: Placebo TPA (N=43) | Week 26 to Week 52: Placebo TPA, Neridronic Acid TPB (N=8) | Week 26 to Week 52: Neridronic Acid TPA (N=39) | Week 26 to Week 52: Neridronic Acid TPA, Neridronic Acid TPB (N=9)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Baseline to Week 26: Placebo TPA (N=51) | Baseline to Week 26: Neridronic Acid TPA (N=48) | Week 26 to Week 52: Placebo TPA (N=43) | Week 26 to Week 52: Placebo TPA, Neridronic Acid TPB (N=8) | Week 26 to Week 52: Neridronic Acid TPA (N=39) | Week 26 to Week 52: Neridronic Acid TPA, Neridronic Acid TPB (N=9)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (12) | 2 (2) | 0 (0) | 2 (5) | 0 (0) | 1 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Acute phase reaction (General disorders) | 5 (6) | 8 (10) | 0 (0) | 2 (9) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complex regional pain syndrome (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (8) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection protozoal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
A pre-specified interim analysis was conducted on pooled primary endpoint data of studies KF7013-04 and KF7013-02 (NCT03530345). The interim analysis indicated futility (neridronate unlikely to be superior to placebo) and both studies were stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any proposed full publication or poster or presentation of the results of this study by the coordinating or other investigator before they are submitted for publication or public disclosure. Neither the sponsor nor the coordinating investigator has the right to prohibit publication or public disclosure. Publication or public disclosure can be postponed for patent purposes.

DOCUMENTS (3):
  • Statistical Analysis Plan: Final-Analysis-KF7013-04 (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT03560986/SAP_000.pdf
  • Statistical Analysis Plan: Pooled-Interim-Analysis-KF7013-02-KF7013-04 (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT03560986/SAP_001.pdf
  • Study Protocol (2018-11-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT03560986/Prot_002.pdf